CLINICAL TRIAL: NCT00196729
Title: A Randomized, Controlled, Open-Label, Multi-National Pilot Study of Thyroid Remnant Ablation Comparing the Safety and Ablation Rate Following 131I Administration Using Thyrogen® Versus the Safety and Ablation Rate Following 131I Administration in the Hypothyroid State
Brief Title: Comparison of the Safety and Successful Ablation of Thyroid Remnant in Post-thyroidectomized Euthyroid Patients (i.e. Patients Administered Thyrogen) Versus Hypothyroid Patients (no Thyrogen) Following 131I Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: THYR00800
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa; Iodine-131

INTERVENTIONS:
Drug: Thyrogen + Radioiodine (131I)

SUMMARY:
This study was conducted in patients with differentiated thyroid cancer who had undergone near-total thyroidectomy. After surgery patients were randomized to one of two methods of performing thyroid remnant ablation (use of radioiodine to remove any remaining thyroid tissue). One group of patients who took thyroid hormone medicine and were euthyroid [i.e. their thyroid stimulating hormone (TSH) levels are normal], and received injections of Thyrogen (0.9 mg daily on two consecutive days) followed by oral radioiodine. The second group of patients did not take thyroid hormone medicine so that they were hypothyroid (i.e. their TSH levels were high), and were given oral radioiodine. All patients received the same amount of radioactive iodine (100 mCi or 3.7 GBq of 131I). Approximately 8 months later, whole body scans were performed on all patients to learn whether the thyroid remnants had been successfully ablated. The safety profile of Thyrogen when used for radioiodine remnant ablation also was assessed. The Quality of Life, the radioiodine uptake and retention into the thyroid bed, as well as radiation exposure to the remainder of the body also were assessed in both groups of patients.

DETAILED DESCRIPTION:
Following a total/near-total thyroidectomy, eligible patients provided written informed consent within 14 days post-surgery. Patients were then randomized to 1 of 2 groups: the Euthyroid or the Hypothyroid group.

Once randomized, patients in the Euthyroid group received thyroid hormone suppression therapy (THST) for 4 weeks. At the end of the fourth week, the patient's TSH level was measured. If the TSH level was < 5 mU/L, Thyrogen (0.9 mg) was administered intramuscularly (IM) once daily (qd) for 2 days. Twenty-four hours following the second dose of Thyrogen, an ablative activity of 131I (100 mCi; 3.7 GBq) was administered. All patients then underwent post-treatment whole-body scanning (WBS) and remnant-neck imaging at 48 hours, at 72 to 96 hours, and at 96 to 168 hours (preferably 120 hours) following ablation. In addition, the study allowed for the option to perform scans at 24 hours and between 144 and 168 hours after ablation. Following the final post-treatment scan, patients in the Euthyroid group continued THST.

Patients randomized to the Hypothyroid Group did not receive THST after randomization. These individuals were monitored for at least 4 weeks or until their TSH was > 25 mU/L. Patients were given an ablative dose of 131I (100 mCi, 3.7 GBq). If the patient's TSH was < 25 mU/L at the end of the fourth week, the patient's TSH was measured again 1 week later. Patients then underwent post-treatment WBS and remnant-neck imaging at 48 hours, at 72 to 96 hours, and at 96 to 168 hours (preferably 120 hours) following ablation. In addition, the study allowed for the option to perform scans at 24 hours and between 144 and 168 hours post ablation. Following the final post-treatment scan, patients in the Hypothyroid group commenced THST.

Eight (± l) months later, patients in both the Euthyroid and Hypothyroid groups received Thyrogen (0.9 mg qd for 2 days) followed by an activity of 131I (4 mCi; 0.15 GBq), in preparation for 48-hour WBS and remnant-neck imaging.

Patients with a negative neck scan (i.e. no visible uptake or, if visible uptake, less than 0.1% uptake in the thyroid bed) 8 (+ 1) months following the 131I treatment were considered successfully ablated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were at least 18 years old (male or female).
* Patients with newly diagnosed differentiated papillary or follicular thyroid carcinoma, including papillary-follicular variant, characterized as "T2, N0 or N1, and M0" or as "T1, N1, and M0".
* Patients with a total or near-total thyroidectomy within 2 weeks prior to enrollment.

Exclusion Criteria:

* see above

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2001-12; Study Completion 2003-09

PRIMARY OUTCOMES:
Use of Thyrogen in euthyroid patients undergoing radioiodine remnant ablation with 100 mCi (3.7 GBq) 131I results in a comparable ablation rate to patients undergoing radioiodine remnant ablation in the hypothyroid state with 100 mCi (3.7 GBq) 131I
Safety profile of Thyrogen when used for radioiodine remnant ablation

SECONDARY OUTCOMES:
QoL in patients treated using Thyrogen
Compare the radioiodine uptake and retention into the thyroid bed in euthyroid patients using Thyrogen and patients treated in the hypothyroid state.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company